CLINICAL TRIAL: NCT06772415
Title: A Phase I Study of Safety, Tolerability, Pharmacokinetics and Preliminary Anti-Tumor Activity of the Oral KIF18A Inhibitor GenSci122 in Participants With Advanced Solid Tumors
Brief Title: A Study to Investigate Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy With GenSci122 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GenSci122-101
Record Dates: First submitted 2025-01-02; First posted 2025-01-13 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: Part 1 Does escalation, Part 2 Dose expansion
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: GenSci122 tablet 50mg; Drug: GenSci122 tablet 250mg

INTERVENTIONS:
Drug: GenSci122 tablet 50mg — Orally Once Daily
Drug: GenSci122 tablet 250mg — Orally Once Daily

SUMMARY:
This is a first-in-human (FIH), multicenter, open-label, phase I study to evaluate the safety, tolerability, PK and preliminary efficacy of GenSci122 in participants with advanced solid tumors. The study consists of 2 parts: Part 1- dose-escalation and Part 2- dose expansion. The primary endpoint of Dose escalation is To assess the safety and tolerability of GenSci122. The primary endpoint of Dose expansion is to evaluate the preliminary anti-tumor activity of GenSci122 in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent and sign the informed consent form (ICF).
2. Male or female participants ≥18 years old at the time of consent.
3. Meeting the requirements of tumor types shown below:

   Dose escalation:

   Participants with a histological or cytological diagnosis of recurrent or metastatic advanced solid tumors who have failed or are intolerant to standard treatment, or have no standard therapy.

   Dose expansion:

   Participants with a histological or cytological diagnosis of recurrent or metastatic advanced solid tumors who have failed or are intolerant to standard treatment, or have no standard therapy.
4. Participants agree to provide fresh or archived tumor tissue as well as corresponding pathological report.
5. Survival expectations are ≥ 12 weeks.
6. Eastern Cooperative Oncology Group performance status (ECOG PS) 0 to 1 (Appendix 1).
7. At least one measurable target lesion
8. Participants with adequate organ function at the time of screening (requiring no blood transfusion, no use of hematopoietic stimulating factor or human albumin or use of drug for correction within 14 days before the first dose)
9. All toxicity related to prior cancer therapies must have resolved to ≤ Grade 1
10. Congestive heart failure (CHF), which must have been ≤ Grade 1 in severity at the time of occurrence and must have resolved completely.
11. Normal QT interval on screening ECG evaluation
12. Participants with a known HIV infection are eligible if the following criteria are met:

    a. Stable on antiretroviral therapy for ≥ 4 weeks before the first dose of GenSci122.

    d. Viral load of < 400 copies per mL at screening. e. CD4+ T-cell count ≥ 350 cells/μL at screening.
13. Hepatitis B virus (HBV) and hepatitis C virus (HCV) test is negative. If participants have active HBV infection: HBV- deoxyribonucleic acid (DNA) must be < 500 IU/mL (or must be < 2500 copy/mL if copy/mL is the only unit available in the study site) and are willing to receive antiviral therapy throughout the study (treatment in accordance with local standard of care, e.g., entecavir); participants with positive HCV ribonucleic acid (RNA) must receive antiviral therapy in accordance with the local standard treatment guideline and have ≤ CTCAE 5.0 Grade 1 elevated hepatic function.
14. Women of childbearing potential (WOCBP) must have a serum pregnancy test negative within 7 days before the first dose of GenSci122. WOCBP must agree to avoid pregnancy during the study and agree to the use 2 effective contraceptive methods (hormonal or barrier method of birth control, or abstinence) before study entry, for the duration of study participation, and in the following 6 months after discontinuation of Gensci122
15. Men with a partner(s) of childbearing potential must take appropriate precautions to avoid fathering a child from screening until 3 months after discontinuation of GenSci122 and to use appropriate barrier contraception or abstinence

Exclusion Criteria:

1. Investigational agent or anticancer therapy within 5 half-lives or 4 weeks (whichever is shorter) before the first dose of GenSci122. In addition, no concurrent investigational anti-cancer therapy is permitted.
2. Major surgery (excluding placement of vascular access) within 4 weeks before the first dose of GenSci122.
3. Radiotherapy within 4 weeks before the first dose of GenSci122. Or participants have not yet recovered from acute effects of radiotherapy to baseline before the first dose of GenSci122.
4. Symptomatic primary central nervous system (CNS) tumor, metastases, leptomeningeal carcinomatosis, or untreated spinal cord compression.
5. Clinically significant active cardiovascular disease or history of myocardial infarction within 6 months before the first dose of GenSci122.
6. Active uncontrolled systemic bacterial, viral, or fungal infection, or serious ongoing intercurrent illness, such as hypertension or diabetes, despite optimal treatment. Screening for chronic conditions is not required.
7. Inability to swallow pills or clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal absorption of GenSci122.
8. Pregnancy or lactation.
9. History of previous cancer, except for squamous cell or basal-cell carcinoma of the skin, or any in situ carcinoma, for which by the date of the first dose of GenSci122, at least 3 years of complete remission and no other treatment is needed or expected during the study period.
10. Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse
11. Allergic to GenSci122 tablet or its components.
12. Any serious illness, uncontrolled inter-current illness, psychiatric illness, or other medical history, including lab results, which in the opinion of investigator or medical monitor would be likely to impact safety or compliance with study requirements or confounds the ability to interpret the data.
13. Has a treatment history of KIF18A inhibitor.
14. Participants with DNA polymerase epsilon (POLE) gene hotspot mutated, or hypermutator phenotype.
15. Other conditions that are not eligible for inclusion based on the investigator's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Dose escalation: Incidence of dose-limiting toxicities (DLTs). | 2 years
Dose expansion: Objective response rate (ORR) evaluated by investigator based on response evaluation criteria in solid tumors version 1.1 (RECIST v1.1). | 3 Years

SECONDARY OUTCOMES:
Incidence and severity of TEAEs. | 3 years
Maximum Plasma Concentration (Cmax) of Gensci122 | 3 years
Time to Maximum Plasma Concentration (Tmax) of Gensci122 | 3 years
Area Under the Plasma Concentration-time Curve (AUC) Over the Dosing Interval for Gensci122 | 3 years
Duration of Response (DOR) | 3 years
Progression-free Survival (PFS) | 3 years
Overall Survival (OS) | 3 years

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The first affiliated hospital of Zhengzhou university, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiang Su Province Hospital, Nanjing, Jiangsu
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - ZhongShan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality